CLINICAL TRIAL: NCT02045199
Title: Efficacy and Safety of V0111 Cream on Open Cracked Heel in Diabetic Patients With Polyneuropathy.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pierre Fabre Medicament (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: V00111 CR 0 02; 2013-A01394-41 (Other: ID RCB Number)
Record Dates: First submitted 2014-01-20; First posted 2014-01-24 (Estimated); Last update posted 2015-04-27 (Estimated); Status verified 2015-04

CONDITIONS: Open Cracked Heel in Diabetic Patients With Polyneuropathy
Keywords: Diabetic Neuropathies; Diabetes Mellitus; Diabetic Foot; Diabetes Complications
MeSH Terms: conditions — Diabetic Neuropathies; Diabetes Mellitus; Diabetic Foot; Diabetes Complications

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- V0111 (Experimental)
  Interventions: Device: Tested product : V0111 cream
- Placebo (Placebo Comparator)
  Interventions: Device: Placebo

INTERVENTIONS:
Device: Tested product : V0111 cream — Application twice a day during 28 days
  Arms: V0111
Device: Placebo — Application twice a day during 28 days
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and the safety of the cream V0111 in the treatment of fissure(s) situated on the heels in diabetic patients with polyneuropathy.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes mellitus with neuropathy,
* Cracked open heel with at least one fissure Grade 2,

Exclusion Criteria:

* Open wound, skin infection, haemorrhagic crack on feet,
* Major static disorder ,
* Ulceration and history of ulceration,
* Active haemorrhagic crack,
* Hyperkeratotic disease
* Diabetic arteriopathy,

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 193 (Actual)
Dates: Start 2014-02; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Complete healing of target fissure on the heel | Day 28
  Comparison of the two treatment groups (verum versus placebo)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Garrigue, MD, Study Director — Pierre Fabre Médicament
Locations (20):
- Belgium (3):
  - Brussels
  - Edegem
  - Liège
- France (17):
  - Angers
  - Bron
  - La Rochelle
  - Laval
  - Mantes-la-Jolie
  - Muret
  - Nanterre
  - Nice
  - Nieuls Sur Mer
  - Paris
  - Pessac
  - Pringy
  - Rillieux Village
  - Saint-Orens-de-Gameville
  - Seysses
  - Suresnes
  - Tiercé